CLINICAL TRIAL: NCT05190653
Title: Early Integration of Palliative and Supportive Care for Patients and Family Caregivers Undergoing Hematopoietic Stem Cell Transplantation or Chimeric Antigen Receptor T-Cell Therapy: A Prospective Pragmatic Randomized Clinical Trial
Brief Title: Early Integration of Palliative and Supportive Care in Cellular Therapy
Acronym: PALS_CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alberta Health Services, Calgary (Other)
Collaborators: Alberta Cancer Foundation (Other); University of Victoria (Other)
Responsible Party: Principal Investigator, Reanne Booker, Principal Investigator, Alberta Health Services, Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 27265
Record Dates: First submitted 2021-12-07; First posted 2022-01-13 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Blood Cancer; Stem Cell Transplant Complications; Chimeric Antigen Receptor T-cell Therapy
Keywords: palliative care; supportive care; quality of life; symptom burden; hematologic malignancies
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Hematologic Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It will not be possible to blind participants or researchers (PC clinicians who will be involved in delivery the intervention) to the intervention but the individual doing the data collection, the research assistant, will be blinded to the randomization allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palliative and Supportive Care Intervention (Experimental): Participants randomized to the intervention arm will meet (either by phone or Zoom contingent upon participant preference) with a palliative care nurse practitioner or palliative care physician. During the first meeting, pre-transplant/CAR T-cell therapy, content will focus on the provision of information and education, including: a description of palliative and supportive care, symptom management, advance care planning, prognostic and illness understanding and treatment expectations, and coping strategies. All subsequent visits will include, at minimum, these topics. All meetings will be audio-recorded using a handheld audio-recorder; the record feature of Zoom will not be utilized. Participants in the intervention arm will meet with a member of the study team (palliative care nurse practitioner or palliative care physician) one to two times weekly, or more frequently if requested by the patient and/or family caregiver, until 3 months post-transplant/CAR T-cell therapy.
  Interventions: Other: Early palliative and supportive care
- Standard Care (No Intervention): Standard care will involve the usual care that patients undergoing HSCT/CAR T-cell therapy would be expected to receive, including palliative care consultation as needed or upon request. Palliative care interventions beyond what are provided in the study will be tracked in both the intervention and the standard care arms.

INTERVENTIONS:
Other: Early palliative and supportive care — The intervention itself will be predominantly the provision of education and information. It is possible that patients in the intervention arm may receive treatment recommendations to help manage symptoms.
  Arms: Palliative and Supportive Care Intervention

SUMMARY:
Research has shown that early palliative care in cancer care is associated with improved symptom management, better prognostic understanding, improved quality of life for patients and family caregivers, and even improved survival. Yet, in spite of the proven benefits of integration of palliative care in oncology, it has been well established that patients with hematologic malignancies and those undergoing cellular therapy (hematopoietic stem cell transplantation (HSCT) and chimeric antigen receptor (CAR) T-cell therapy) do not routinely receive palliative care. Most of the published research on the early integration of palliative care in oncology describes studies that have involved patients with solid tumours. To date, only one randomized trial examining the impact of integrated palliative care among patients undergoing HSCT has been published and there have been no studies examining the impact of integrated palliative care for patients undergoing CAR T-cell therapy. The American Society of Clinical Oncology recommends early palliative care for patients with advanced cancers or for those with high symptom burden. Patients with blood cancers experience high symptom burden and in the last 30 days of life, compared to patients with solid tumours, patients with blood cancers are more likely to die in hospital, have more intensive care unit admissions, have prolonged hospitalizations (>14 days), and pass away in an acute care facility. There is an urgent need to proactively address suffering throughout cellular therapy trajectories, even before treatment starts, so that patients and caregivers are not inevitably waiting for symptoms to arise before they can be addressed and to optimize quality of life for patients undergoing transplant as well as their family caregivers.

PALS_CT will compare early palliative care to standard care for patients and their family caregivers undergoing HSCT or CAR T-cell therapy for blood cancers.

DETAILED DESCRIPTION:
Problem: patients undergoing HSCT and CAR T-cell therapy experience high symptom burden (physical, psychological, spiritual), lack illness and prognostic understanding (which can adversely impact medical decision making). Research has found that patients with blood cancers experience poor end-of-life (EOL) quality indicators such as disease-directed therapy in the weeks before death, emergency room visits in the weeks before death, intensive care unit (ICU) admissions near the EOL, low rates of hospice use, and dying in hospital. Family caregivers (CGs) of patients undergoing HSCT and CAR T-cell therapy experience impaired QOL, physical and psychosocial concerns, and have expressed that their needs have not been adequately addressed by care teams. Palliative care, with its multidisciplinary approach and focus on improving QOL from a holistic perspective, can help reduce symptom burden and improve QOL, improve illness and prognostic understanding, and improve EOL care for patients undergoing HSCT and CAR T-cell therapy and their family CGs. This trial will assess the effectiveness of early PC in improving QOL for patients and their family CGs undergoing HSCT or CAR T-cell therapy for hematological malignancies.

Objectives The objectives for this study were developed after extensive review of the literature as well as were informed by preliminary data derived from an ongoing qualitative study that sought the perspectives of patients, family CGs, and clinicians regarding the integration of PC in HSCT.

Objective 1: To examine the impact of an outpatient PC intervention on patient-reported QOL for patients undergoing HSCT or CAR T-cell therapy Hypothesis: patients randomized to the PC intervention will report greater improvement in QOL at 1-month post-HSCT/CAR T-cell therapy and at 3 months post-HSCT/CAR T-cell therapy compared to patients receiving standard care.

Objective 2: To examine the impact of an outpatient PC intervention on symptoms at 2 weeks, 1 month, and 3 months post-HSCT/CAR T-cell therapy for patients undergoing HSCT/CAR T-cell therapy Hypothesis: patients randomized to the PC intervention will report a greater reduction in physical symptoms at 2 weeks, 1 month, and 3 months post-HSCT/CAR T-cell therapy compared to patients receiving standard care

Objective 3: To examine the impact of an outpatient PC intervention on family CG QOL at 1 month and 3 months post-HSCT/CAR T-cell therapy for CGs of patients undergoing HSCT/CAR T-cell therapy Hypothesis: family CGs of patients randomized to the PC intervention will report greater improvement in QOL compared to family CGs of patients receiving standard care

Objective 4: To examine the impact of an outpatient PC intervention on patient and family CG understanding of prognosis.

Hypothesis: patients and family CGs randomized to the PC intervention will report more accurate prognostic understanding compared to those receiving standard care

Exploratory objective 1: To evaluate whether an outpatient PC intervention is associated with overall survival at 1 and 5 years post-study enrolment.

Methods This is a prospective pragmatic randomized clinical trial to evaluate the effectiveness of an outpatient PC intervention integrated with standard care compared to standard care alone in 152 patients undergoing HSCT or CAR T-cell therapy. Randomization will be stratified by type of treatment: autologous transplant, allogeneic transplant, or CAR T-cell therapy. A pragmatic approach was selected given the desire to assess the effectiveness of integrating early PC in HSCT/CAR T-cell therapy. Previous studies have examined the efficacy of PC in oncology in patients with advanced cancer. This study will build the work of El-Jawahri et al. who studied the impact of inpatient PC on patients undergoing HSCT with the main difference being that participants will be recruited in the outpatient setting and the intervention will be delivered in the outpatient setting. Selected outcomes have been chosen as they are congruent with patient, family CG and clinician perspectives, based upon the qualitative study that was undertaken by the PI (R Booker) in 2020-2021.

Data Collection Participants will be emailed a secure link for the questionnaires. Data from questionnaires will be collected electronically using Research Electronic Data Capture (REDCap). Email reminders will be sent to participants to remind them to complete the surveys and if necessary, a research assistant will contact patients and family CGs to provide reminders to complete the surveys.

Following randomization, participants (patients and family CGs) will be asked to complete baseline questionnaires and demographic information (such as age, gender, diagnosis, urban/rural residence, religious affiliation, highest level of education, main CG (for patients), main source of support (for family CGs) will be collected via REDCap. The next evaluation will occur during the second week following HSCT or CAR T-cell therapy. For participants undergoing autologous HSCT or CAR T-cell therapy (and their family CGs), the second evaluation will occur on day +5 (with a 48-hour window). For participants undergoing allogeneic HSCT (and their family CGs), the second evaluation will occur on day +8 (with a 72-hour window). These time points were chosen based upon the study conducted by El-Jawahri et al. who indicated they selected the time points to coincide with the peak of severity in symptoms based upon the type of transplant being performed. All patients and family CGs will also complete questionnaires at 1 and 3 months post HSCT/CAR T-cell therapy. Data collection will be done remotely, with links to questionnaires sent via email completed via REDCap. As part of the consent process, participants will be asked if they would consider completing questionnaires at 6-12 months post-HSCT/CAR T-cell therapy. Patient participants will also be asked if they consent to the researchers accessing their medical charts until 5 years post-HSCT/CAR T-cell therapy in order to collect disease and treatment information.

Data Analysis Exclusive intention-to-treat (ITT) analysis may not be aligned with patient-centered outcomes and as such, this study will use both ITT and per protocol analyses. For any imbalances between the intervention and control groups, sensitivity analyses while be conducted and g-methods will be used to adjust for confounders that may vary over time. As per the revised CONSORT guidelines for reporting parallel-group randomized trials, the investigators will collect and report the reasons for participants lost to follow-up as well as the reasons why any participants' data were excluded from analysis.

Analysis Plan Primary Outcome To assess the primary outcome of the study, difference in QOL, as measured by the MQOL-E, between the intervention group and the standard care group will be compared. Because QOL will be assessed at multiple time points, area under the curve (AUC) will be used to calculate a summary score for each patient. Assessing multiple domains over time increases the possibility of Type I error. In particular, because it is expected that patient trajectories of QOL will be non-linear, AUC seems more appropriate than using specific time points as the latter may underestimate or overestimate treatment differences. Summary scores will be averaged across all patients in both the intervention and standard care arms and differences between the groups will be assessed using t-tests. The summary profiles for patients will be presented in graphical form for the MQOL and FACT-BMT.

Analysis Plan - Secondary Outcomes Family CG QOL will be analyzed using AUC and comparing the two groups using t-tests. For patient symptom burden, as measured by the ESAS, symptom scores will be tracked over time for each patient. An overall summary score for the ESAS will not be used given the diversity of symptoms assessed by the ESAS as well as the possibility that patients can add another symptom or concern to the tool. The latter would mean that there could be different symptoms being reported amongst participants, thereby making it difficult to compare groups. Patient and family CG prognostic understanding will be assessed using t-tests to compare the intervention group and standard care group at two time points, pre-HSCT/CAR T-cell therapy and at 3 months post-HSCT/CAR T-cell therapy.

ELIGIBILITY:
Inclusion Criteria - Patients

* Clinical diagnosis of hematologic malignancy with scheduled hematopoietic stem cell transplantation or chimeric antigen receptor (CAR) T-cell therapy
* Ability to speak, read, and understand English or, be able to complete questionnaires with minimal assistance required from an interpreter

Inclusion Criteria - Family Caregivers

* Family caregivers of patients with a clinical diagnosis of hematologic malignancy with scheduled hematopoietic stem cell transplantation or chimeric antigen receptor (CAR) T-cell therapy
* A spouse, relative, or friend, identified by the patient, who either lives with the patient or has in-person contact with the patient at least twice per week. Only one family CG per patient will be asked to participate.
* Ability to speak, read, and understand English or willing to complete questionnaires with minimal assistance required from an interpreter

Exclusion Criteria - Patients

* Patients undergoing HSCT for a non-malignant hematologic condition
* Inability to provide informed consent

Exclusion Criterion - Family Caregivers

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2025-04-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient quality of life | 3 months
  The primary outcome of the study, QOL, will be assessed using the McGill Quality of Life Questionnaire - Expanded (MQOL-E) summary score of QOL monthly for a period of three months. The MQOL-E consists of 21 items with possible scores of 0 to 10 for each item. The higher the score, the better the QOL. The trajectories of QOL will be evaluated rather than looking at change in scores as it is anticipated that there will be significant fluctuation in QOL scores over time. The Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) will also be used to measure QOL. The FACT-BMT is more specific to BMT and may capture issues that are unique to BMT. The FACT-BMT consists of 47 items; a 5-point Likert-type scale is used for item. The total score ranges from 0-196 and higher scores indicate better QOL.

SECONDARY OUTCOMES:
Patient symptom burden | 3 months
  The Edmonton Symptom Assessment System (ESAS) is a validated scale that assesses symptom burden in patients with cancer. While several iterations of the ESAS are available, this study will use the ESAS-revised (ESAS-r) which includes 10 items scored using a numeric rating scale, where 0=no symptom and 10=worst symptom. The ESAS assesses physical symptoms (pain, fatigue, nausea, drowsiness, dyspnea, loss of appetite), emotional symptoms (anxiety and depression), and well-being. Individual patient scores will be tracked over time to assess the trajectory of symptom burden.
Patient and family caregiver prognostic understanding | 3 months
  The Perception of Treatment and Prognosis Questionnaire (PTPQ) is 10 item self-report questionnaire that assesses patients' beliefs about the likelihood of cure, the importance and helpfulness of knowing about prognosis, the primary goal of cancer treatment, the preferences for information about treatment, and the satisfaction with quality of information provided regarding prognosis and treatment. Items on the questionnaire are scored individually with statements about the degree to which the patient agrees with each item. Patients and CGs will complete the PTPQ pre-HSCT/CAR T-cell therapy and at 3 months post HSCT/CAR T-cell therapy.
Family caregiver quality of life | 3 months
  The Quality of Life in Life-Threatening Illness - Family carer version 2 (QOLLTI-F v2) will be used to assess CG QOL. The QOLLTI-Fv2 is a 17-item questionnaire that includes seven subscales that assess the following domains: environment, patient condition, the CG's own state, quality of care, relationships, and financial worries. In addition, there is a single item that pertains to overall QOL. Items on the QOLLTI-Fv2 are ranked from 0-10 (total possible score ranges from 0-170), where higher scores are associated with better QOL. Caregivers in both the intervention and standard care arms will complete the QOLLTI-Fv2 pre-HSCT/CAR T-cell therapy, and at 2-weeks, 1-month, and 3-months post-HSCT/CAR T-cell therapy.

OTHER OUTCOMES:
1 year overall survival | 1 year
  Patient survival at 1 year post-study enrolment
5 year overall survival | 5 years
  Patient survival at 5 years post-study enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Reanne Booker, PhD(c), Principal Investigator — AHS Calgary
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Jawahri A, LeBlanc T, VanDusen H, Traeger L, Greer JA, Pirl WF, Jackson VA, Telles J, Rhodes A, Spitzer TR, McAfee S, Chen YA, Lee SS, Temel JS. Effect of Inpatient Palliative Care on Quality of Life 2 Weeks After Hematopoietic Stem Cell Transplantation: A Randomized Clinical Trial. JAMA. 2016 Nov 22;316(20):2094-2103. doi: 10.1001/jama.2016.16786. PMID 27893130
- [Background] Hui D, Didwaniya N, Vidal M, Shin SH, Chisholm G, Roquemore J, Bruera E. Quality of end-of-life care in patients with hematologic malignancies: a retrospective cohort study. Cancer. 2014 May 15;120(10):1572-8. doi: 10.1002/cncr.28614. Epub 2014 Feb 18. PMID 24549743
- [Background] Hui D, Hannon BL, Zimmermann C, Bruera E. Improving patient and caregiver outcomes in oncology: Team-based, timely, and targeted palliative care. CA Cancer J Clin. 2018 Sep;68(5):356-376. doi: 10.3322/caac.21490. Epub 2018 Sep 13. PMID 30277572
- [Background] Kaasa S, Loge JH, Aapro M, Albreht T, Anderson R, Bruera E, Brunelli C, Caraceni A, Cervantes A, Currow DC, Deliens L, Fallon M, Gomez-Batiste X, Grotmol KS, Hannon B, Haugen DF, Higginson IJ, Hjermstad MJ, Hui D, Jordan K, Kurita GP, Larkin PJ, Miccinesi G, Nauck F, Pribakovic R, Rodin G, Sjogren P, Stone P, Zimmermann C, Lundeby T. Integration of oncology and palliative care: a Lancet Oncology Commission. Lancet Oncol. 2018 Nov;19(11):e588-e653. doi: 10.1016/S1470-2045(18)30415-7. Epub 2018 Oct 18. PMID 30344075
- [Background] Temel JS, Greer JA, El-Jawahri A, Pirl WF, Park ER, Jackson VA, Back AL, Kamdar M, Jacobsen J, Chittenden EH, Rinaldi SP, Gallagher ER, Eusebio JR, Li Z, Muzikansky A, Ryan DP. Effects of Early Integrated Palliative Care in Patients With Lung and GI Cancer: A Randomized Clinical Trial. J Clin Oncol. 2017 Mar 10;35(8):834-841. doi: 10.1200/JCO.2016.70.5046. Epub 2016 Dec 28. PMID 28029308
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Gray TF, Temel JS, El-Jawahri A. Illness and prognostic understanding in patients with hematologic malignancies. Blood Rev. 2021 Jan;45:100692. doi: 10.1016/j.blre.2020.100692. Epub 2020 Apr 6. PMID 32284227
- [Background] Hochman MJ, Yu Y, Wolf SP, Samsa GP, Kamal AH, LeBlanc TW. Comparing the Palliative Care Needs of Patients With Hematologic and Solid Malignancies. J Pain Symptom Manage. 2018 Jan;55(1):82-88.e1. doi: 10.1016/j.jpainsymman.2017.08.030. Epub 2017 Sep 5. PMID 28887271
- [Background] Ferrell BR, Temel JS, Temin S, Alesi ER, Balboni TA, Basch EM, Firn JI, Paice JA, Peppercorn JM, Phillips T, Stovall EL, Zimmermann C, Smith TJ. Integration of Palliative Care Into Standard Oncology Care: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Jan;35(1):96-112. doi: 10.1200/JCO.2016.70.1474. Epub 2016 Oct 28. PMID 28034065
- [Background] El-Jawahri A, Nelson AM, Gray TF, Lee SJ, LeBlanc TW. Palliative and End-of-Life Care for Patients With Hematologic Malignancies. J Clin Oncol. 2020 Mar 20;38(9):944-953. doi: 10.1200/JCO.18.02386. Epub 2020 Feb 5. PMID 32023164
- [Background] El-Jawahri A, Traeger L, Kuzmuk K, Eusebio J, Vandusen H, Keenan T, Shin J, Gallagher ER, Greer JA, Pirl WF, Jackson VA, Ballen KK, Spitzer TR, Graubert TA, McAfee S, Dey B, Chen YB, Temel JS. Prognostic understanding, quality of life and mood in patients undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2015 Aug;50(8):1119-24. doi: 10.1038/bmt.2015.113. Epub 2015 May 11. PMID 25961772